CLINICAL TRIAL: NCT06189261
Title: Feasibility and Acceptability of a Holistic Needs Assessment Intervention Employing Patient-reported Outcome Measures (PROMs) to Support Newly Diagnosed Patients With Malignant Melanoma
Brief Title: Holistic Needs Assessments in Patients With Melanoma
Status: Completed | Type: Observational
Sponsor: University of Surrey (Other)
Responsible Party: Sponsor
Other Study IDs: RE4090
Record Dates: First submitted 2016-03-01; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Melanoma; Unsatisfied Needs
Keywords: Supportive care; Unsatisfied needs; Melanoma; Holistic assessment; Patient-reported outcomes; PROMs
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with stage 1/2 malignant melanoma: During the study, two intervention consultations will take place 1 and 3 months after the initial clinical team meeting, where each participant's case will be discussed. At the start of each intervention consultation, patients will be asked to complete the intervention questionnaire. The recorded information will be passed to their nurse specialist, who will identify the participant's needs and offer tailored advice and support to meet these needs. Throughout the study, participants will also be asked to complete a set of questionnaires in the clinic (months 1 and 3) or at home (months 2 and 4) to explore potential effects of the intervention.
  Interventions: Other: Holistic needs assessment based on the use of patient-reported outcome measures

INTERVENTIONS:
Other: Holistic needs assessment based on the use of patient-reported outcome measures — During the study, two intervention consultations will take place 1 and 3 months after the initial clinical team meeting, where each participant's case will be discussed. At the start of each intervention consultation, participants will be asked to complete the intervention patient-reported outcome measure (i.e. Distress Thermometer and Problem Checklist, and Supportive Care Needs Survey-Melanoma Module). The recorded information will be passed to their nurse specialist, who will identify the participant's needs and offer tailored advice and support to meet these needs.

SUMMARY:
This study will assess whether a needs assessment/management intervention for patients with malignant melanoma is achievable, reasonable, realistic and of value to patients with malignant melanoma and health professionals involved in their care.

The study will also explore what the levels of patients' unmet needs are, whether unmet needs change over time, and what the potential effects of the intervention may be on patients' unmet needs, symptom severity, self-confidence in dealing with the illness, wellbeing, and satisfaction with the care received.

In this study, the investigators will involve skin cancer nurse specialists, who will be asked to use an 'intervention questionnaire' to offer a needs assessment/management intervention to 30 people newly diagnosed with malignant melanoma. The investigators have used information from the literature to select the most appropriate 'intervention questionnaire' for this patient population.

Each consenting patient (i.e. participant) will be expected to participate in the study over 4 months. During the study, two intervention consultations will take place 1 and 3 months after the initial clinical team meeting, where each participant's case will be discussed. At the start of each intervention consultation, participants will be asked to complete the intervention questionnaire. The recorded information will be passed to their nurse specialist, who will identify the participant's needs and offer tailored advice and support to meet these needs.

Throughout the study, participants will also be asked to complete a set of questionnaires in the clinic (months 1 and 3) or at home (months 2 and 4) to explore potential effects of the intervention. A study evaluation form will be used at month 4 to collect participants' and health professionals' views on the intervention and how it was delivered. Face-to-face interviews will take place at the end of the study to explore participants' (a subset of 10 people) and health professionals' experiences with the intervention.

DETAILED DESCRIPTION:
no additional detail, study has ended

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of malignant melanoma Stage I or II regardless of tumour thickness.
* Within 1 month post-initial diagnosis following a MDT meeting.
* Aged 18 years or over.
* Deemed by a member of the MDT to be physically and psychologically fit to participate.
* Able to read and write English.
* Able to provide written informed consent.

Exclusion Criteria:

* Patients not meeting the afore-mentioned criteria will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A convenience sample of up to 30 newly diagnosed patients with malignant melanoma will be recruited from out-patient clinics at one NHS board in Scotland.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-02; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Feasibility of intervention | Baseline to end of study, a total of 9 months
  Data on patient availability/recruitment, time and resource requirements, missing data, patient retention will be recorded and analysed.
Acceptability of intervention | Baseline to end of study, a total of 9 months
  Data on adherence to intervention, perceived burden, timing of intervention will be collected through interviews with participants and health professionals.

SECONDARY OUTCOMES:
Supportive Care Needs Survey-Short Form 34 (SCNS-SF34) | Baseline (first consultation), 1 month post-baseline (follow-up), 2 months post-baseline (second consultation), 3 months post-baseline (follow-up)
  no additional detail, study completed
Quality of Life (Functional Assessment of Cancer Therapy - Melanoma (FACT-M) | Baseline (first consultation), 1 month post-baseline (follow-up), 2 months post-baseline (second consultation), 3 months post-baseline (follow-up)
  no additional detail, study completed
Self-efficacy (Communication and Attitudinal Self-Efficacy scale - Cancer (CASE-Cancer) | Baseline (first consultation), 1 month post-baseline (follow-up), 2 months post-baseline (second consultation), 3 months post-baseline (follow-up)
  no additional detail, study completed
Experiences of care (Patient Satisfaction with Cancer Care questionnaire (PSCC) | 1 month post-baseline (follow-up), 3 months post-baseline (follow-up
  no additional detail, study completed
Edmonton Symptom Assessment System (ESAS) | Baseline (first consultation), 1 month post-baseline (follow-up), 2 months post-baseline (second consultation), 3 months post-baseline (follow-up)
  no additional detail, study completed
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core30 (EORTC QLQ-C30) and EORTC Melanoma-38 (MEL-38) | Baseline (first consultation), 3 months post-baseline (follow-up)
  no additional detail, study completed

CONTACTS AND LOCATIONS:
Overall Officials: Roma Maguire, PhD, Principal Investigator — University of Surrey
Locations (1):
- Monklands Hospital, NHS Lanarkshire, Glasgow, Lanarkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised individual participant data (IPD) collected as part of this project will be used in publications and presentations following the end of the study. In addition, anonymised IPD will be shared with colleagues from the European Organisation for Research and Treatment of Cancer (EORTC) Melanoma research group to aid the psychometric development of the new Melanoma module of the EORTC Quality of Life Questionnaire-Core 30 (QLQ-C30) questionnaire. Written patient consent will be sought before any data are shared with the above-mentioned group.